## Impact of the Gut Microbiome on Health Impacts of Haskap Berries

Dr. Mary Miles

NCT #: 2024-1417-FCR

November 5, 2024

## Statistical Analysis:

Analysis of blood markers will be done in the latest version of R Studio available at the time. Linear models and analysis of variances assessments will be used to compare responses before and after the 8-week intervention. Anthropometric measures relevant to variables, like visceral adiposity and inflammation, will be added as potential covariates. Metabolomic analysis of before and after intervention samples will be analyzed using the latest version of Metaboanalyst at the time and the latest version of R Studio available at the time. Stool samples will be analyzed via 16s sequencing to determine the microbial community in each participant. R studio will be used to analyze the changes to microbial diversity over the course of the intervention and correlate blood marker findings with the microbial communities present.